CLINICAL TRIAL: NCT06104410
Title: Optimization of Fractionation Schedules of Heel Spur Radiotherapy: Monocentric Prospective Randomized Open-label Trial
Brief Title: Optimization of Fractionation Schedules of Heel Spur Radiotherapy Prospective Randomized Open-label Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Masaryk Memorial Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NU22-10-00479
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Heel Spur
MeSH Terms: conditions — Heel Spur

STUDY DESIGN:
Intervention Model Description: The trial is designed as binary outcome parallel group non-inferiority trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (standard fractionated dose): Groups A-B (Active Comparator): Arm A contains of 2 groups. Group A: Total dose of 6 Gy in 4 single fractions of 1.5 Gy applied twice weekly (most commonly used regimen, considered standard arm in this trial) Group B: Total dose of 3 Gy in 2 single fractions of 1.5 Gy applied twice weekly
  Interventions: Radiation: Standard fractioned dose
- Arm B (experimental single dose): Groups C-F (Experimental): Arm B contains of four groups. Group C: Total dose of 0.5 Gy in 1 single fractions of 0.5 Gy Group D: Total dose of 1 Gy in 1 single fractions of 1 Gy Group E: Total dose of 1.5 Gy in 1 single fractions of 1.5 Gy Group F: Total dose of 2 Gy in 1 single fractions of 2 Gy
  Interventions: Radiation: Experimental single dose

INTERVENTIONS:
Radiation: Standard fractioned dose — Total dose of 6 Gy in 2 or 4 single fractions of 1.5 Gy applied twice weekly.
  Arms: Arm A (standard fractionated dose): Groups A-B
Radiation: Experimental single dose — Total dose of 0.5 Gy, 1Gy, 1.5 or 2Gy in 1 single fraction.
  Arms: Arm B (experimental single dose): Groups C-F

SUMMARY:
About 26 000 patients are treated per year with radiotherapy for non-malignant diseases in the Czech Republic, majority of them with heel spur syndrome which prevalence ranges from 8-10% in the general population. Heel spur represents important socioeconomic as well as health care issue. Radiotherapy by orthovoltage X-ray belongs to standard conservative treatment methods with proven antiinflammatory effect. Nevertheless, with increasing incidence of cancer, it may be assumed that availability of radiotherapy service for heel spur patients will be further limited including limitations related to potential pandemic or other emergency situation. This represents upcoming unmet clinical need, where alternative approaches with dramatically abbreviated fractionation schedules are needed in order to keep availability as well as effectivity of heel spur (and other non-malignant disorders) radiotherapy.

The aim to presented single institutional prospective randomized open-lable clinical trial is to evaluate low dose radiotherapy delivered in single fraction manner in the treatment of heel spur syndrome.

The project aims to design a randomized trial that compared fractionated and single fraction radiotherapy (non-inferiority). Patients will be randomized into 6 groups according to the total dose, total of 966 patients will be enrolled. The primary objective is to compare Calcaneodynia sum score at 3 months after radiotherapy between fractionated vs. single fraction radiotherapy.

DETAILED DESCRIPTION:
Purpose/Objective The aim of this study is to optimize the fractionation schedules for radiotherapy in the treatment of heel spurs (HSS, plantar fasciitis) through a prospective randomized open-label trial conducted at Department of Radiation Oncology at Masaryk Memorial Cancer Institute Brno (MMCI). Low-dose external beam radiotherapy (LD-EBRT), known for its anti-inflammatory effect, offers effective pain relief for HSS patients. Currently, the standard LD-EBRT regimen consists of six fractions of 1 Gray (Gy) administered twice weekly, resulting in a total dose of 6 Gy. This study posits the hypothesis that very low total doses of orthovoltage radiotherapy, delivered in a single fraction, may provide pain relief comparable to that achieved with higher doses of fractionated radiotherapy. The primary goal of this research is to determine whether one-day irradiation (a single fraction) is non-inferior to fractionated radiotherapy over a three-month period in terms of pain relief for HSS patients. This study was supported by grant of the Ministry of Health of the Czech Republic AZV NU22-10-00479. All patients signed informed consent.

Material/Methods After completing the enrollment process and filling out the SF-36 questionnaire, as well as the Calcaneodynia score (CS) and visual analogue pain score (VAS) forms, patients (pts) meeting specific inclusion criteria (being over 40 years old, having a diagnosed painful unilateral plantar HSS for at least six months, and being suitable for HSS radiotherapy), and fulfilling the main exclusion criteria (having no prior history of radiotherapy for heel spur, no corticosteroid local application in the four weeks leading up to radiotherapy, no systemic rheumatic or collagen vascular diseases, lymphatic edema of the lower limb, or prior trauma and surgery on the ipsilateral foot), were randomized into six groups based on the total dose of radiotherapy. Patients in these groups received a total dose of 6 Gy in 4 fractions of 1.5 Gy twice weekly (arm A), a total dose of 3 Gy in 2 fractions of 1.5 Gy twice weekly (arm B), a single fraction of 0.5 Gy (arm C), a single fraction of 1.0 Gy (arm D), a single fraction of 1.5 Gy (arm E), and a single fraction of 2 Gy (arm F), respectively. The regimen in arm A (6 Gy in 4 fractions) is commonly used in MMCI and considered as the standard arm. In the event of inadequate pain relief, reirradiation was performed with a total dose of 6 Gy in 4 fractions of 1.5 Gy twice weekly after a waiting period of three months in any of the aforementioned groups.

ELIGIBILITY:
All patients referred to medical attention for non-malignant radiotherapy at the Department of Radiation oncology, Masaryk Memorial Cancer Institute (MMCI), will be screened for eligibility, and if all inclusion/exclusion criteria are met, they will be invited to participate in the present study.

Inclusion Criteria:

* 1) Patients aged over 40 years who have been diagnosed clinically and radiologically to be suffering from a painful unilateral plantar heel spur for at least six months,
* 2) indication to heel spur radiotherapy,
* 3) 40 years or older patient, good performance status (Karnofsky index ≥ 70),
* 4) exclusion of other local diseases by the orthopaedic surgeon,
* 5) willingness of the patient to provide telephone or email contact to maintain follow up.

Exclusion Criteria:

* 1) Prior radiotherapy of heel spur (even if prior radiotherapy was performed on the contralateral heel spur because of possible bias given patient's expectations and experiences related to previous radiotherapy,
* 2) corticosteroid local application during last 4 weeks prior to planned radiotherapy,
* 3) rheumatic or vascular diseases, lymphatic edema of lower limb,
* 4) former trauma or surgery of ipsilateral foot,
* 5) any systemic illness (collagen vascular diseases) or unstable medical condition that might pose additional risk for performance of radiotherapy including claustrophobia or jactation,
* 6) any other factors that, in the opinion of the site investigators, would interfere with adherence to study requirements,
* 7) pregnancy or breastfeeding,
* 8) inability or unwillingness of subject to sign written informed consent.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority of single fraction radiotherapy of heel spur | 44 months
  Comparison of 2 arms in 3 months after radiotherapy.Follow-up examinations consist of personal examination,questionnaire survey.Calcaneodynia sum score (100=free of symptoms, 0=very intense symptoms) is calculated by evaluation of Pain symptoms (up to 30 points),Use of appliances (up to 15 points),Professional activities (up to 20 points),Daily/leisure activities (up to 15 points) and Gaint/limp (up to 20 points). Complete pain relief will be assumed if patients will be completely free of pain and regained full ability to walk and function well.Insufficient pain relief will be assumed,if the patient's subjective evaluation (VAS score) of improvement of pain will be less than 80% or if the temporal pattern of clinical response will be unsatisfactory (ie, response will be delayed >3 months or there will be need for second radiotherapy course.Skin toxicity will be evaluated according Common Terminology Criteria for Adverse Events (CTCAE) v5. VAS and SF36 are described in Outcome 4.

SECONDARY OUTCOMES:
Comparison of different single fraction radiotherapy prescription | 44 months
  Comparison of Calcaneodynia sum score at 3 months after radiotherapy between different single fraction radiotherapy prescription. Calcaneodynia sum score (100 = free of symptoms, 0 = very intense symptoms) is calculated by evaluation of Pain symptoms (up to 30 points), Use of appliances (up to 15 points), Professional activities (up to 20 points), Daily/leisure activities (up to 15 points) and Gaint/limp (up to 20 points).
Comparison of the need for reirradiation till 1 year after radiotherapy between fractionated vs. single fraction radiotherapy | 44 months
  To compare the need for reirradiation till 1 year after radiotherapy between fractionated vs.
  single fraction radiotherapy. To compare the need of reirradiation till 1 year after radiotherapy between different single fraction radiotherapy prescription. Evaluated simply by keeping score of patients returning for irradiation till 1 year after radiotherapy.
Comparison of quality of life and VAS score at 1.5, 3, 6, 9 and 12 months and Calcaneodynia sum score at 1.5, 6, 9 and 12 months between fractionated vs. single fraction radiotherapy and between different single fractions radiotherapy prescription. | 44 months
  Visual analogue scale (VAS) score is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain." (0 = no pain, 100 = maximum imaginable pain intensity).SF-36 questionnaire score taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions and single item that provides an indication of perceived change in health. High values indicates good quality of life.
Evaluation of individual (not sum) parts of Calcaneodynia score and individual domains of quality of life | 44 months
  Evaluation of individual (not sum) parts of Calcaneodynia score and individual domains of quality of life as per outcome 1,2 and 4. Calcaneodynia score form is attached in separate file in this project proposal. Sum score (100 = free of symptoms, 0 = very intense symptoms) is calculated by evaluation of Pain symptoms (up to 30 points), Use of appliances (up to 15 points), Professional activities (up to 20 points), Daily/leisure activities (up to 15 points) and Gaint/limp (up to 20 points).
Analysis of the heel spur radiotherapy techniques in Czechia | 44 months
  Conducting a questionnaire survey analyzing the technique of heel spur radiotherapy at individual workplaces performing this type of treatment in Czechia. The questionnaires will be conducted by Masaryk Memorial Cancer Institute and sent to other facilities in Czechia. Results will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Slampa, prof. MD, Principal Investigator — Masaryk Memorial Cancer Institute
Locations (1):
- Masaryk Memorial Cancer Institute, Brno, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dufek V, Zackova H, Kotik L, Horakova I. RESULTS OF CZECH NATIONAL STUDY OF RADIATION EXPOSURE FROM RADIOTHERAPY OF NON-MALIGNANT DISEASES, IN PARTICULAR OF HEEL SPURS. Radiat Prot Dosimetry. 2019 Dec 31;186(2-3):386-390. doi: 10.1093/rpd/ncz237. PMID 31840171
- [Background] Buchbinder R. Clinical practice. Plantar fasciitis. N Engl J Med. 2004 May 20;350(21):2159-66. doi: 10.1056/NEJMcp032745. No abstract available. PMID 15152061
- [Background] DeMaio M, Paine R, Mangine RE, Drez D Jr. Plantar fasciitis. Orthopedics. 1993 Oct;16(10):1153-63. doi: 10.3928/0147-7447-19931001-13. No abstract available. PMID 8255812
- [Background] Heyd R, Tselis N, Ackermann H, Roddiger SJ, Zamboglou N. Radiation therapy for painful heel spurs: results of a prospective randomized study. Strahlenther Onkol. 2007 Jan;183(1):3-9. doi: 10.1007/s00066-007-1589-1. PMID 17225939
- [Background] Barrett SJ, O'Malley R. Plantar fasciitis and other causes of heel pain. Am Fam Physician. 1999 Apr 15;59(8):2200-6. PMID 10221305
- [Background] Kriz J, Seegenschmiedt HM, Bartels A, Micke O, Muecke R, Schaefer U, Haverkamp U, Eich HT. Updated strategies in the treatment of benign diseases-a patterns of care study of the german cooperative group on benign diseases. Adv Radiat Oncol. 2018 Feb 26;3(3):240-244. doi: 10.1016/j.adro.2018.02.008. eCollection 2018 Jul-Sep. PMID 30197936
- [Background] Crawford F, Thomson C. Interventions for treating plantar heel pain. Cochrane Database Syst Rev. 2003;(3):CD000416. doi: 10.1002/14651858.CD000416. PMID 12917892
- [Background] Seegenschmiedt MH, Keilholz L, Katalinic A, Stecken A, Sauer R. Heel spur: radiation therapy for refractory pain--results with three treatment concepts. Radiology. 1996 Jul;200(1):271-6. doi: 10.1148/radiology.200.1.8657925.
- [Background] Seegenschmiedt MH, Keilholz L, Stecken A, Katalinic A, Sauer R. [Radiotherapy of plantar heel spurs: indications, technique, clinical results at different dose concepts]. Strahlenther Onkol. 1996 Jul;172(7):376-83. German. PMID 8693404
- [Background] Trott KR. Therapeutic effects of low radiation doses. Strahlenther Onkol. 1994 Jan;170(1):1-12. PMID 8303572
- [Background] Bentzen SM. Radiation therapy: intensity modulated, image guided, biologically optimized and evidence based. Radiother Oncol. 2005 Dec;77(3):227-30. doi: 10.1016/j.radonc.2005.11.001. Epub 2005 Nov 21. No abstract available. PMID 16300846
- [Background] Kern P, Keilholz L, Forster C, Seegenschmiedt MH, Sauer R, Herrmann M. In vitro apoptosis in peripheral blood mononuclear cells induced by low-dose radiotherapy displays a discontinuous dose-dependence. Int J Radiat Biol. 1999 Aug;75(8):995-1003. doi: 10.1080/095530099139755. PMID 10465365
- [Background] Kern PM, Keilholz L, Forster C, Hallmann R, Herrmann M, Seegenschmiedt MH. Low-dose radiotherapy selectively reduces adhesion of peripheral blood mononuclear cells to endothelium in vitro. Radiother Oncol. 2000 Mar;54(3):273-82. doi: 10.1016/s0167-8140(00)00141-9. PMID 10738086
- [Background] Niewald M, Seegenschmiedt MH, Micke O, Graeber S, Muecke R, Schaefer V, Scheid C, Fleckenstein J, Licht N, Ruebe C; German Cooperative Group on Radiotherapy for Benign Diseases (GCGBD) of the German Society for Radiation Oncology (DEGRO). Randomized, multicenter trial on the effect of radiation therapy on plantar fasciitis (painful heel spur) comparing a standard dose with a very low dose: mature results after 12 months' follow-up. Int J Radiat Oncol Biol Phys. 2012 Nov 15;84(4):e455-62. doi: 10.1016/j.ijrobp.2012.06.022. Epub 2012 Jul 25. PMID 22836057
- [Background] Ott OJ, Jeremias C, Gaipl US, Frey B, Schmidt M, Fietkau R. Radiotherapy for benign calcaneodynia: long-term results of the Erlangen Dose Optimization (EDO) trial. Strahlenther Onkol. 2014 Jul;190(7):671-5. doi: 10.1007/s00066-014-0618-0. Epub 2014 Mar 26. PMID 24668250
- [Background] Rowe CR, Sakellarides HT, Freeman PA, Sorbie C. Fractures of the Os Calcis: A Long-Term Follow-up Study of 146 Patients. JAMA. 1963;184(12):920-923. doi:10.1001/jama.1963.03700250056007